CLINICAL TRIAL: NCT02217085
Title: Determining True Colorectal Polyp Resection Adequacy: Correlation of Endoscopic Margins With Histopathologic Margins
Brief Title: Colorectal Polyp Resection Adequacy
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: RSA-RTSC 2014
Record Dates: First submitted 2014-07-14; First posted 2014-08-15 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Polyp Resection Adequacy
Keywords: Colorectal Cancer Screening; Colon Cancer Screening; Polyps; Colonoscopy
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Polyp margins will be biopsied and retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to determine the best way to ensure that polyps are completely removed by evaluating the borders of the removed polyp. If a polyp is found that meets the size requirements for the study, the investigators will take extra biopsies of the margin to determine if there is any abnormal tissue or cancer at these borders.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80

Exclusion Criteria:

* Coagulopathy (international normalized ratio >2)
* Inflammatory bowel disease or other active colitides
* Polyps of index colonoscopy that were felt not to be completely resected or pedunculated
* Familial adenomatous polyposis or hereditary polyposis
* Potential hereditary cancer syndrome (Lynch Syndrome)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 40 to 80 who are undergoing screening or surveillance colonoscopy for colorectal adenomatous polyps.
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2014-05; Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
The incomplete resection rates in polyps from Group 1 (clear margins) versus Group 2 (positive margins). | Between 3-6 months
  Define the frequency of free margins versus margins that have dysplasia to the cautery site in snare polypectomy. A free margin is defined as uninvolved or normal mucosa extending to the cautery margin at the polypectomy stalk.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States